CLINICAL TRIAL: NCT06972849
Title: BabyCCINO: Caffeine Citrate to Improve Neonatal Outcomes. A Neonatal Domain Within PLATIPUS.
Brief Title: Caffeine Citrate to Improve Neonatal Outcomes.
Acronym: BabyCCINO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P-N01-BabyCCINO
Record Dates: First submitted 2025-04-27; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-04

CONDITIONS: Apnea of Prematurity
Keywords: Preterm infant; Apnea of Prematurity; Apnoea of Prematurity; Caffeine citrate
MeSH Terms: conditions — Apnea; Premature Birth | interventions — caffeine citrate

STUDY DESIGN:
Intervention Model Description: BabyCCINO is a domain within the PLATIPUS adaptive platform trial (NCT06461429).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All parties will be blinded to the assigned intervention arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Caffeine citrate 40mg (Active Comparator): Dose and frequency 40mg/kg load and 20mg/kg maintenance daily, as long as clinically indicated.
  Administration Loading dose: 2mL/kg loading dose of study drug, either IV or enterally, administered at <72 hours of life, followed by Maintenance dose: 1mL/kg maintenance dose given daily, either IV or enterally, commenced 24 hours after loading dose.
  Interventions: Drug: Caffeine citrate
- Caffeine citrate 30mg (Active Comparator): Dose and frequency 30 mg/kg load and 15mg/kg maintenance daily, as long as clinically indicated.
  Administration Loading dose: 2mL/kg loading dose of study drug, either IV or enterally, administered at <72 hours of life, followed by Maintenance dose: 1mL/kg maintenance dose given daily, either IV or enterally, commenced 24 hours after loading dose.
  Interventions: Drug: Caffeine citrate
- Caffeine citrate 20mg (Active Comparator): Dose and frequency 20mg/kg load and 10mg/kg maintenance daily, as long as clinically indicated.
  Administration Loading dose: 2mL/kg loading dose of study drug, either IV or enterally, administered at <72 hours of life, followed by Maintenance dose: 1mL/kg maintenance dose given daily, either IV or enterally, commenced 24 hours after loading dose.
  Interventions: Drug: Caffeine citrate

INTERVENTIONS:
Drug: Caffeine citrate — Clinically indicated for apnea of prematurity.
  Other Names: Cafcit

SUMMARY:
The goal of this clinical trial to learn what dose/s of caffeine citrate works to treat preterm born babies who have episodes where they stop breathing. It will also learn about the safety of different doses of caffeine citrate for the variety of preterm-born babies that are prescribed this.

The main question it aims to answer is: Which dose is the optimal dose of caffeine citrate for very preterm babies to prevent short-term death and disease?

Researchers will compare three different doses of caffeine citrate, which are already used in clinical practice to treat breathing stoppages in preterm babies, to see which dose works best. No placebo will be used.

Participants will be given a 'loading' dose of caffeine citrate <72 hours of life, and a smaller 'maintenance' dose once a day, for as long as the baby needs this.

This trial will be undertaken as part of the PLATIPUS trial (NCT06461429).

DETAILED DESCRIPTION:
The BabyCCINO trial will compare the efficacy and safety of a higher, medium or lower-dose caffeine regimen in very preterm infants. It is a neonatal domain within the PLATIPUS adaptive platform trial (NCT06461429).

Apnoea of prematurity, which causes repeated episodes of low oxygen saturation, affects virtually all extremely preterm infants born <28 weeks' gestation and more than half of those born 28-31 weeks' gestation. Apnoeic events are associated with poorer neurodevelopmental outcomes in infancy. Some very preterm infants also require mechanical ventilation due to apnoea, with an associated risk of bronchopulmonary dysplasia (BPD), the chronic lung disease of prematurity diagnosed at 36 weeks' post-menstrual age (PMA).

Caffeine is one of the most commonly prescribed drugs in neonatal medicine and reduces apnoea of prematurity. The largest trial of caffeine in very preterm infants, the Caffeine for Apnea of Prematurity (CAP) trial, found that caffeine improves important short-term respiratory outcomes and longer-term brain development compared with placebo. There is evidence from small clinical trials of more benefit from higher dose caffeine than that used in the CAP trial, however, potential side effects include jitteriness, tachycardia and feed intolerance. A higher rate of cerebellar haemorrhage was also reported in one small trial in infants who received a higher loading dose of 80 mg/kg, along with a trend to higher seizure burden however, a Cochrane review did not identify any adverse effects of higher-dose caffeine.

BabyCCINO will compare three dosing regimens routinely prescribed in Australia and Aotearoa New Zealand and assess health outcomes for infants who receive these.

Very preterm infants born <32 weeks' gestation will be randomly assigned to receive either

* 40mg/kg loading dose and 20mg/kg daily maintenance
* 30 mg/kg loading dose and 15mg/kg daily maintenance, or
* 20mg/kg loading dose and 10mg/kg daily maintenance.

Health outcomes will be assessed using the PLATIPUS Ordinal Outcome Scale, at 42 weeks' postmenstrual age or discharge home, whichever is earliest.

ELIGIBILITY:
PLATFORM ELIGIBILITY

Participants must meet all core PLATIPUS platform inclusion criteria:

* Born before 37 weeks gestation
* Receiving pregnancy care at a participating site (hospital) at the time of eligibility assessment and
* Meet eligibility criteria for one or more platform domains.

Participants will be excluded from participation if they meet any core PLATIPUS platform exclusion criteria:

* (Parent) Inability to consent for their infant, unless a domain-level waiver of consent is deemed appropriate.
* Perinatal death is deemed to be imminent and inevitable during the next 24 hours (at time of screening), including if neonatal intensive care is not being provided to the infant.

Infants who meet ALL of the core platform inclusion criteria and none of the exclusion criteria will be considered for BabyCCINO-specific eligibility.

BabyCCINO-SPECIFIC ELIGIBILITY

Platform-eligible participants must meet all BabyCCINO-specific inclusion criteria:

1. Very preterm infants born <32 weeks' gestation
2. <72 hours old
3. Very preterm infants born at <32 weeks' gestation, <72 hours of age, with any clinical indication for commencing caffeine, as determined by the treating clinician, including:

   * Prevention or treatment of apnoea
   * Facilitating extubation from mechanical ventilation
   * Prevention of BPD
   * For longer-term benefit.

Participants will be excluded from participation if they meet any BabyCCINO-specific exclusion criteria:

1. Prior treatment with caffeine, other methylxanthines, or doxapram
2. Major congenital anomalies: major congenital cardiac disease (not including patent ductus arteriosus or isolated atrial/ventricular septal defects), major gastrointestinal malformations, congenital diaphragmatic hernia, known genetic syndromes, known brain malformations
3. Death considered to be imminent in the next 24 hours, or intensive care not going to be offered or continued
4. Pre-existing tachyarrhythmia (e.g., antenatal or postnatal supraventricular tachycardia)
5. Pre-existing seizures
6. No parental/caregiver consent or not satisfying the principles and criteria for waiver with consent to continue, as approved in the relevant jurisdiction

Platform-eligible participants who meet all BabyCCINO-specific inclusion criteria and none of the BabyCCINO-specific exclusion criteria will be eligible to participate in BabyCCINO.

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3900 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2050-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants who progress by at least one level higher on the PLATIPUS Ordinal Outcome Scale | At any time prior to 42 weeks' postmenstrual age or first discharge home from hospital (whichever is earlier)
  The PLATIPUS-Ordinal Outcome Scale ranks the most severe core short-term infant health outcome in the specified time frame.
  Levels 1-15: 1= Well, liveborn infant; 2= Neonatal unit admission for <48 hours; 3= Neonatal unit admission for >/= 48 hours; 4= Non-invasive respiratory support or oxygen therapy for ≥ 4 hours & < 5 days; 5= Non-invasive respiratory support or oxygen therapy >/= 5 days; 6= Mechanical ventilation via endotracheal tube for ≥ 4 hours & <7 days; 7= Mechanical ventilation via endotracheal tube for >/=7 days; 8= Moderate respiratory morbidity; 9=Necrotising enterocolitis AND/OR Sepsis; 10= Severe Respiratory Morbidity; 11= Major Surgery; 12= Brain Injury; 13= TWO of severe respiratory morbidity OR major surgery OR brain injury; 14= Severe respiratory morbidity & major surgery & brain injury; 15 = Death.

SECONDARY OUTCOMES:
Number of infants with moderate respiratory morbidity (as per the primary outcome) | At any time prior to 42 weeks' postmenstrual age or first discharge home from hospital (whichever is earlier).
  Number of infants meeting the PLATIPUS-Ordinal Outcome Scale definition of 'moderate respiratory morbidity'.
Number of infants with severe respiratory morbidity (as per the primary outcome) | At any time prior to 42 weeks' postmenstrual age or first discharge home from hospital (whichever is earlier).
  Number of infants meeting the PLATIPUS-Ordinal Outcome Scale definition of 'severe respiratory morbidity'.
Duration of any positive pressure ventilation, in days | From first date and time (any mode), to final date and time (any mode), up to 42 weeks' postmenstrual age or first discharge home from hospital (whichever is earlier)
  Any positive pressure ventilation (mechanical ventilation, non-invasive positive pressure ventilation, continuous positive airway pressure or nasal high-flow therapy), in days (in survivors to 42 weeks' PMA or first discharge home from hospital, whichever is sooner).
Duration of mechanical ventilation, in days | From start date and time, to end date and time, up to 42 weeks' postmenstrual age or first discharge home from hospital (whichever is earlier)
  Mechanical ventilation, in days (in survivors to 42 weeks' PMA or first discharge home from hospital, whichever is sooner).
Number of infants with patent ductus arteriosus treated with medication or surgery | At any time prior to 42 weeks' postmenstrual age or first discharge home from hospital (whichever is earlier)
  Number of infants with patent ductus arteriosus treated with medication or surgery.
Number of infants with retinopathy of prematurity receiving intraocular or laser treatment | At any time prior to 42 weeks' postmenstrual age or first discharge home from hospital (whichever is earlier)
  Number of infants with retinopathy of prematurity receiving intraocular or laser treatment.
Number of infants treated with postnatal systemic corticosteroids for preterm lung disease | At any time prior to 42 weeks' postmenstrual age or first discharge home from hospital (whichever is earlier)
  Number of infants treated with postnatal systemic corticosteroids for preterm lung disease.
Number of infants with presumed caffeine side-effects | At any time prior to 42 weeks' postmenstrual age or first discharge home from hospital (whichever is earlier)
  Number of infants with presumed caffeine side-effects, where the treating clinician has reduced the dose or ceased caffeine.

OTHER OUTCOMES:
Core Secondary Outcome 1: Number of participants in each, individual component of the primary outcome. | At any time prior to 42 weeks' postmenstrual age or first discharge home from hospital (whichever is earlier)
  The PLATIPUS-Ordinal Outcome Scale (primary outcome) ranks the most severe core short-term infant health outcome in the specified time frame.
  Levels 1-15: 1= Well, liveborn infant; 2= Neonatal unit admission for <48 hours; 3= Neonatal unit admission for >/= 48 hours; 4= Non-invasive respiratory support or oxygen therapy for ≥ 4 hours & < 5 days; 5= Non-invasive respiratory support or oxygen therapy >/= 5 days; 6= Mechanical ventilation via endotracheal tube for ≥ 4 hours & <7 days; 7= Mechanical ventilation via endotracheal tube for >/=7 days; 8= Moderate respiratory morbidity; 9=Necrotising enterocolitis AND/OR Sepsis; 10= Severe Respiratory Morbidity; 11= Major Surgery; 12= Brain Injury; 13= TWO of severe respiratory morbidity OR major surgery OR brain injury; 14= Severe respiratory morbidity & major surgery & brain injury; 15 = Death.
Core Secondary Outcome 2: Infant growth measures | At 42 weeks postmenstrual age or first discharge home from hospital (whichever is earliest).
  Head circumference (measured in cms), weight (measured in gms), length (measured in cms) and growth z-score will be calculated at 42 weeks postmenstrual age, or first discharge home from hospital (whichever is earliest)
Core Secondary Outcome 3: Total duration of first hospitalisation (birth admission) | From date of birth to date first discharged home from hospital
  Duration of first hospitalisation, measured in days.
Core Secondary Outcome 4: Rate of (any) breastmilk feeding at 42 weeks postmenstrual age, or on the day of first discharge home from hospital. | On the day of 42+0 weeks postmenstrual age or first discharge home from hospital (whichever is earliest)
  Any breastmilk feeding (any mode - breast, bottle or tube) at 42 weeks postmenstrual age, or on the day of first discharge home from hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Brett Manley, MBChB PhD, Principal Investigator — University of Melbourne

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will align with PLATIPUS (NCT06461429) policy. Version 1, Apr-2024
  Once data unblinding no longer compromises the integrity of the trial, a de-identified data set collected for the analysis of domains within PLATIPUS will be made available.
  Conditions:
  1. All domains in which the participant is co-enrolled are closed to recruitment* (*Where one or more domains in which a participant is co-enrolled are not yet closed to recruitment, the participant's data may be provided, without the treatment code, to prevent unblinding in unfinished domains).
  2. Primary domain conclusions/analyses have been published, AND
  3. The 2-year follow-up of participants within the domain/s of interest is/are complete.
  Supporting materials (Core Protocol, Domain-Specific Appendices, Data Dictionaries and Domain-Specific Statistical Analysis Plans) will be available.
  Contact: University of Melbourne - info@platipustrial.org.
Supporting Information: Study Protocol, SAP
Time Frame: This is estimated to be approximately six months following the completion of the two-year follow-up of domain participants.
Access Criteria: To be determined. Access requests will be subject to review by trial subcommittees. The Trial Steering Committee will approve or disapprove requests. A Data Transfer Agreement and Authorship Agreement signed by relevant parties and evidence of ethical approval will be required.